CLINICAL TRIAL: NCT05032287
Title: Medical Expulsive Therapy Post-SWL For Renal Stones. A Randomized Trial
Brief Title: Medical Expulsive Therapy Post-SWL For Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MET SWL
Record Dates: First submitted 2021-08-25; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Urologic Diseases; Urolithiasis; Stone, Kidney
MeSH Terms: conditions — Urologic Diseases; Urolithiasis; Kidney Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tamsulosin (Active Comparator): tamsulosin 0.4 mg once daily
  Interventions: Drug: Tamsulosin
- Placeb (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin 0.4 mg once daily
  Arms: tamsulosin
Drug: Placebo — Placebo once daily
  Arms: Placeb

SUMMARY:
To evaluate the efficacy and stone free rate of placebo versus tamsulosin as medical expulsive therapy post-SWL in patients with renal stone less than 20 mm

ELIGIBILITY:
Inclusion Criteria:

* Renal stone ≤ 20 mm.
* Lower calyceal stone ≤ 15 mm

Exclusion Criteria:

* Women with known or suspected pregnancy or breastfeeding.
* History of alpa-blockers (more than 7 days prior to study participation)
* History of ureteral stricture
* Multiple (that is more than 2) stones
* Stone in solitary kidney (either anatomically or functionally).
* Presence of urinary sepsis.
* Estimated glomerular filtration rate < 30 ml/min
* Contraindication or allergy to tamsulosin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Stone free rate defined as patient free of any stone residual | at 3 months
  assessed by Non-contrast Computed Tomography of Urinary Tract (NCCT-UT)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt